CLINICAL TRIAL: NCT03373578
Title: Comparison of the Preterm Newborn Sleep With and Without the Use of Earmuffs During the "Quiet Time" in a Neonatal Unit
Brief Title: Earing Protectors Influence on Newborns Preterm Sleep Pattern
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Mavilde da Luz Gonçalves Pedreira, Escola Paulista de Enfermagem, Federal University of São Paulo
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: Unifesp003
Record Dates: First submitted 2014-08-07; First posted 2017-12-14 (Actual); Last update posted 2017-12-14 (Actual); Status verified 2014-08

CONDITIONS: Sleep
Keywords: sleep;; Infant, Premature;; Polysomnography;; Ear Protective Devices
MeSH Terms: conditions — Premature Birth | interventions — Ear Protective Devices

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- earmuffs (Active Comparator): Preterm newborns with earmuffs during the Quiet time
  Interventions: Device: earmuffs
- control (No Intervention): Preterm newborns without earmuffs during de Quiet time

INTERVENTIONS:
Device: earmuffs — to compare the neonate's sleep with and without earmuffs during Quiet time at the NICU
  Arms: earmuffs

SUMMARY:
Preterm newborn sleep deprivation due to medical interventions and environmental characteristics of the Neonatal Intermediate Care Unit (NICU) can increase morbidity and developmental deleterious effects. The aim of this study is to test the effect of earmuffs on sleep pattern of preterm neonates. Prospective, randomized, controlled, crossover study conducted in NICU of two teaching hospitals from São Paulo, Brazil. The effect of earmuffs use was analyzed through polysomnography measurement during four "Quiet times" periods. It was also analyzed sleep related variables during 24 hours of the day. Preterm newborns characteristics and clinical characteristics were also analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Preterm Newborns inside the incubator;
* Preterm Newborns clinically stable;
* Preterm Newborns with no change in hearing screening test;
* Preterm Newborns current weight between 1200 and 2000g.

Exclusion Criteria:

* Preterm Newborns in phototherapy;
* Preterm Newborns in use of invasive mechanical ventilation and noninvasive;
* Preterm Newborns with any type of congenital malformation;
* Preterm Newborns with periventricular hemorrhage grades II, III and IV;
* Preterm Newborns that received Central Nervous System depressant medication and sedative opioid analgesics in the last 24 hours;
* Preterm Newborns using corticoids;
* Preterm Newborn whose mother has a history of illicit drug use during pregnancy

Max Age: 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Sleep period | 4 periods of Quiet time (60 minutes)
  categorized as the total time of sleep measured by polysomnography

SECONDARY OUTCOMES:
sleep pattern according to environmental variables | 4 periods of Quiet time (60 minutes)
  polysomnographic records and clinical environmental variables

CONTACTS AND LOCATIONS:
Overall Officials: Eliana M Pinheiro, phD, Study Director — Federal University of São Paulo; Mônica H Sato, MSc, Principal Investigator — Federal University of São Paulo; Mavilde LG Pedreira, phD, Study Director — Federal University of São Paulo; Ariane M Avelar, phD, Study Chair — Federal University of São Paulo
Locations (1):
- Federal Uiversity of São Paulo, São Paulo, Brazil